CLINICAL TRIAL: NCT03572114
Title: Imaging Neuromelanin and Iron in Dystonia/Parkinsonism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0075; IRAS ID 243171 (Other: UCL R&D)
Record Dates: First submitted 2018-02-08; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Sporadic Dystonia; Dystonia, Familial; Parkinson Disease, Juvenile; Neurodegeneration With Brain Iron Accumulation 5; Mitochondrial Diseases
MeSH Terms: conditions — Dystonic Disorders; Parkinsonian Disorders; Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Sporadic Dystonia: 3 Tesla MRI Burke-Fahn-Marsden Dystonia Rating scale MDS-United Parkinsons Disease Rating Scale, Part III Beck Depression Inventory MoCA: Montreal Cognitive Assessment
  Interventions: Diagnostic Test: 3Tesla MRI; Behavioral: Burke-Fahn-Marsden Dystonia Rating scale; Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III; Behavioral: Beck Depression Inventory; Behavioral: MoCA: Montreal Cognitive Assessment:
- Familial Dystonia: 3 Tesla MRI Burke-Fahn-Marsden Dystonia Rating scale MDS-United Parkinsons Disease Rating Scale, Part III Beck Depression Inventory MoCA: Montreal Cognitive Assessment
  Interventions: Diagnostic Test: 3Tesla MRI; Behavioral: Burke-Fahn-Marsden Dystonia Rating scale; Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III; Behavioral: Beck Depression Inventory; Behavioral: MoCA: Montreal Cognitive Assessment:
- Parkinson´s disease, juvenile: 3 Tesla MRI Burke-Fahn-Marsden Dystonia Rating scale MDS-United Parkinsons Disease Rating Scale, Part III Beck Depression Inventory MoCA: Montreal Cognitive Assessment
  Interventions: Diagnostic Test: 3Tesla MRI; Behavioral: Burke-Fahn-Marsden Dystonia Rating scale; Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III; Behavioral: Beck Depression Inventory; Behavioral: MoCA: Montreal Cognitive Assessment:
- Neurodegeneration with brain iron acc.: 3 Tesla MRI Burke-Fahn-Marsden Dystonia Rating scale MDS-United Parkinsons Disease Rating Scale, Part III Beck Depression Inventory MoCA: Montreal Cognitive Assessment
  Interventions: Diagnostic Test: 3Tesla MRI; Behavioral: Burke-Fahn-Marsden Dystonia Rating scale; Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III; Behavioral: Beck Depression Inventory; Behavioral: MoCA: Montreal Cognitive Assessment:
- mitochondrial disease: 3 Tesla MRI Burke-Fahn-Marsden Dystonia Rating scale MDS-United Parkinsons Disease Rating Scale, Part III Beck Depression Inventory MoCA: Montreal Cognitive Assessment
  Interventions: Diagnostic Test: 3Tesla MRI; Behavioral: Burke-Fahn-Marsden Dystonia Rating scale; Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III; Behavioral: Beck Depression Inventory; Behavioral: MoCA: Montreal Cognitive Assessment:
- Healthy Controls: 3 Tesla MRI Burke-Fahn-Marsden Dystonia Rating scale MDS-United Parkinsons Disease Rating Scale, Part III Beck Depression Inventory MoCA: Montreal Cognitive Assessment
  Interventions: Diagnostic Test: 3Tesla MRI; Behavioral: Burke-Fahn-Marsden Dystonia Rating scale; Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III; Behavioral: Beck Depression Inventory; Behavioral: MoCA: Montreal Cognitive Assessment:

INTERVENTIONS:
Diagnostic Test: 3Tesla MRI — 1. A previously validated multi-parameter mapping protocol sensitive to neuromelanin and iron content
  2. Iron mapping and micro-bleed detection: QSM (quantitative susceptibility mapping), a fully flow-compensated, susceptibility-weighted gradient-echo sequence (5 minutes).
  3. 1-mm isotropic anatomical MPRAGE (magnetization-prepared rapid gradient-echo)
  4. conventional FLAIR sequence
Behavioral: Burke-Fahn-Marsden Dystonia Rating scale — internationally standardized examination/quantification of dystonia
Behavioral: MDS-United Parkinsons Disease Rating Scale, Part III — most recent, internationally standardized examination/quantification of bradykinesia / rigidity according to the Movement Disorder Society
Behavioral: Beck Depression Inventory — internationally standardized examination to quantify traits of anxiety and depression
Behavioral: MoCA: Montreal Cognitive Assessment: — internationally standardized examination to quantify cognition, frequently used in studies of dystonia and parkinsonism

SUMMARY:
To generate pilot data to investigate the potential to use in vivo iron- and neuromelanin-quantification as imaging tools for the diagnostic evaluation of movement disorders with predominant dystonia / parkinsonism. To this end we are planning to compare the MR imaging neuromelanin and iron-pattern and content in midbrain, striatum and further brain structures in clinically similar entities and respective, sex- and age-matched healthy controls.

DETAILED DESCRIPTION:
Iron- or Neuromelanin-sensitive MR-imaging has not been consistently applied to the study of syndromes presenting with predominant dystonia/parkinsonism yet. We are planning to study the following groups, as they can often be very difficult to be distinguished from PD and in particular young-onset PD, on clinical grounds only:

* Dopa-responsive dystonia (DRD) can present similar to young-onset PD, but carries a completely different prognosis, necessitating different treatment requirements due to fundamentally different underlying physiology.
* Sporadic and Inherited dystonias (i.e. due to TorsinA (DYT1) and other gene mutations) often present with dystonia, particularly affecting the leg, which is clinically indistinguishable from young-onset PD.
* Young-onset PD, i.e. PD presenting with motor symptoms before 45 years of age, caused by a familiar gene mutation (PARKIN, Pink, DJ-1, PLA2G6, FBX07, ATP13A2, VPS13C, RAB39B, Lubag), often presents with predominant dystonia, particularly with leg-onset.
* NBIAs present with dystonia/parkinsonism: while basal ganglia iron accumulation is a known hallmark feature of the condition [3], the characteristics of neuromelanin regulation are unknown.
* Mitochondrial disease presenting with dystonia / parkinsonism (such as for example Leigh syndrome due to mutations in the Surf-1 gene or mutations m.3243A>G or POLG) [4]
* Respective age- and sex-matched healthy controls This study is designed to produce pilot data on these disease entities. By potentially accelerating the diagnostic process and identification of disease entities, neurologists might be able to deliver more selective and dedicated treatment.

Furthermore, combining Neuromelanin- and iron-specific imaging will offer the possibility to study the condition- specific dynamics of iron homeostasis in these rare conditions.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of parkinsonism and/or dystonia due to
* dopa-responsive dystonia
* sporadic or inherited/genetic dystonia
* young-onset Parkinson's disease
* NBIA
* Mitochondrial disease

  * OR healthy controls
  * 18 to 60 years of age
  * able to give informed consent

Exclusion Criteria:

* Inability to tolerate 35min in an MRI machine
* Participated in a clinical drug trial up to 28 days before inclusion into the present study
* Contra-indications to 3T MRI on MRI safety grounds, such as presence of contra-indicated medical implants, as according to the established routine operating procedures for clinical MRI in the Lysholm Department of Neuroradiology at the National Hospital for Neurology and Neurosurgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients from the National Hospital of Neurology, Queen Square, movement disorder outpatient clinic;
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
neuromelanin content | up to 8 weeks
  absolute amount of neuromelanin in midbrain, striatum and other areas of the brain

SECONDARY OUTCOMES:
neuromelanin association | up to 8 weeks
  correlate neuromelanin quantification with demographic and clinical details
iron association | up to 8 weeks
  correlate neuromelanin quantification with demographic and clinical details
Iron content | up to 8 weeks
  absolute amount of iron in midbrain, striatum and other areas of the brain

CONTACTS AND LOCATIONS:
Overall Officials: Bhatia P Kailash, MD, DM, FRCP, Principal Investigator — UCL, Institute of Neurology, Sobell Department

IPD SHARING:
Plan to Share IPD: No